CLINICAL TRIAL: NCT06938568
Title: Personalized Physical Back Training Program to Improve Physical Functioning in People With Non-specific Low Back Pain
Acronym: LIFDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudio Perret (Other)
Responsible Party: Sponsor-Investigator, Claudio Perret, Prof. Dr. Claudio Perret, Universität Luzern
Organization: Universität Luzern (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-01285; 63674 (Other Grant/Funding Number: Stiftung Universität Luzern)
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Exercise Therapy; Low Back Pain
Keywords: Physical Functioning; Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized back exercises (Experimental): The study intervention is a 12-week personalized physical back training program. It consists of six to eight exercises selected from a predefined set by a physical therapist or medical doctor. These exercises are selected through a clinical reasoning process, i.e., they are tailored and problem-oriented, based on the results of a clinical assessment.
  Interventions: Other: Personalized back exercises
- Non-personalized back exercises (Active Comparator): The active control intervention is a 12-week non-personalized physical back training program. It consists of six to eight exercises selected from a predefined set by a physical therapist or medical doctor. These exercises are not selected through a clinical reasoning process, i.e., they are neither tailored nor problem-oriented nor based on the results of a clinical assessment.
  Interventions: Other: Non-personalized back exercises

INTERVENTIONS:
Other: Personalized back exercises — The study intervention is a 12-week personalized physical back training program. It consists of six to eight exercises selected from a predefined set by a physical therapist or medical doctor. These exercises are selected through a clinical reasoning process, i.e., they are tailored and problem-oriented, based on the results of a clinical assessment.
  An initial one-on-one training session will take place to familiarize participants with the back training program, corresponding to the first week's session of the 12-week intervention period. During the 12-week intervention period, the training comprises one supervised group session per week, lasting 30 minutes, along with three individual unsupervised sessions, each lasting 10-15 minutes. Our procedures ensures that both participants and instructors are blinded to the group allocation, allowing both groups to train together (e.g., mixed training groups).
  Arms: Personalized back exercises
Other: Non-personalized back exercises — The active control intervention is a 12-week non-personalized physical back training program. It consists of six to eight exercises selected from a predefined set by a physical therapist or medical doctor. These exercises are not selected through a clinical reasoning process, i.e., they are neither tailored nor problem-oriented nor based on the results of a clinical assessment.
  An initial one-on-one training session will take place to familiarize participants with the back training program, corresponding to the first week's session of the 12-week intervention period. During the 12-week intervention period, the training comprises one supervised group session per week, lasting 30 minutes, along with three individual unsupervised sessions, each lasting 10-15 minutes. Our procedures ensures that both participants and instructors are blinded to the group allocation, allowing both groups to train together (e.g., mixed training groups).
  Arms: Non-personalized back exercises

SUMMARY:
Personalized medicine and individualized therapeutic approaches are prominent in current research. But are these approaches also effective for treating non-specific low back pain (NSLBP)? NSLBP is one of the most common musculoskeletal issues, which can impair physical well-being, reduce the quality of life, and limit physical functioning. Additionally, it contributes to substantial direct and indirect healthcare costs, such as frequent doctor visits and work absences. Despite NSLBP being a significant burden for both individuals and society, effective alleviation methods remain unclear. The investigators' research project therefore aims to investigate whether personalized therapy, specifically a personalized physical back training program, can effectively address NSLBP. Within the context of NSLBP, the investigators' specific aim is to improve physical functioning as this outcome is considered relevant from all perspectives, including those of patients, clinical professionals, researchers, and guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Access to the University Sports of the Lucerne Universities (i.e., students, employees, alumni, subscribers)
* NSLBP for at least 6 weeks
* Activity limiting NSLBP (at least one activity with a PSFS Score of ≤ 50/100 on a scale from 0 = unable to perform due to NSLBP to 100 = able to perform at the same level as before NSLBP)
* Age between 18 and 65 years
* Understand the German language
* Willing to participate in the study
* Written informed consent

Exclusion Criteria:

* Specific LBP
* Red flags associated with any serious pathology or specific LBP,
* Being on a waiting list for or less than 12 months post any surgery of the lower back
* Pregnancy or given birth within the last 12 months
* Diagnosed central neurological disease
* Not allowed to exercise
* Participant in the feasibility study
* Expecting to be absent for more than 2 weeks during the intervention period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Self-rated physical functioning | Baseline to 12 weeks
  Change in Patient-Specific Functional Scale (PSFS), most bothersome activity. Range from 0 (unable to perform due to NSLBP) to 100 (able to perform at the same level as before NSLBP)

SECONDARY OUTCOMES:
Self-rated physical functioning | Baseline to 4, 8, and 24 weeks
  Change in Patient-Specific Functional Scale (PSFS), most bothersome activity. Range from 0 (unable to perform due to NSLBP) to 100 (able to perform at the same level as before NSLBP)
Self-rated physical functioning (RMDQ) | Baseline to 4, 8, 12, and 24 weeks
  Change in Roland Morris Disability Questionnaire (RMDQ). Range from 0 (no disability) to 24 (maximum disability).
Health-related quality of life (EQ-VAS) | Baseline to 4, 8, 12, and 24 weeks
  Change in EQ Visual Analogue Scale (EQ-VAS). Range from 0 (lowest health-related quality of life) to 100 (highest health-related quality of life).
Health-related quality of life (EQ-5D-5L) | Baseline to 4, 8, 12, and 24 weeks
  Change in 5-Level EuroQoL5D version (EQ-5D-5L). Range from 0 (lowest health-related quality of life) to 1 (highest health-related quality of life).
Pain intensity (NRS) | Baseline to 4, 8, 12, and 24 weeks
  Change in pain intensity (11-point Numeric Rating Scale, NRS). Range from 0 (no pain) to 10 (pain as bad as you can imagine). Recall period: 7 days.
Safety outcome | During the 12 week intervention period
  Number of serious adverse events (SAE) and adverse events (AE) that are deemed possibly, probably, or definitely related to the intervention (according to our protocol and ClinO, Art. 63, Switzerland).

OTHER OUTCOMES:
Pain frequency | Baseline to 4, 8, 12, and 24 weeks
  Change in number of episodes with NSLBP. Numerically, with 0 = minimum. Recall period: 7 days.
Pain duration | Baseline to 4, 8, 12, and 24 weeks
  Change in pain duration (e.g., average duration of an episode of NSLBP within the last 7 days). In minutes, hours, or days, with 0 = minimum. Recall period: 7 days.
Pain interference (PEG) | Baseline to 4, 8, 12, and 24 weeks
  Change in Pain, Enjoyment, and General Activity (PEG) 3-Item Scale. Range from 0 (no pain; does not interfere) to 10 (pain as bad as you can imagine; completely interferes). Recall period: 7 days.
NSLBP-related work productivity loss | Baseline to 4, 8, 12, and 24 weeks
  Change in Work Productivity and Activity Impairment Questionnaire (WPAI). Percentages, with 0%=no work productivity loss.
Participant satisfaction | At 4, 8, 12, and 24 weeks
  Participant satisfaction (e.g., 1. I am satisfied with the training program I received. 2. I am satisfied with the result of the training program). 4-point Likert scale (strongly agree, agree, disagree, strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Perret, PhD, Principal Investigator — University of Lucerne, University Research Centre Health and Society
Locations (1):
- University of Lucerne, Faculty of Health Sciences and Medicine, University Research Centre Health and Society, Lucerne, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that the investigators will make encrypted individual participant data (IPD) available via a data repository and, additionally, upon reasonable request to the Principal Investigator. In both cases, only data from participants who have provided informed consent for data sharing will be made available.
Time Frame: It is anticipated that the data will be made available as soon as possible after the completion of the study and will remain accessible for at least 10 years.
Access Criteria: Access to the data will be granted in accordance with the criteria of the repository and/or publisher.